CLINICAL TRIAL: NCT04393610
Title: Magnesium Sulphate Versus Fentanyl: Effects on the Quality of Bier Block: Double Blind Placebo Controlled Trial
Brief Title: Improving Quality of Bier Block
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RAGAA AHMED HERDAN, Associate Professor of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Quality IVRA
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Analgesia
Keywords: Magnesium sulphate; Fentanyl; Bier block
MeSH Terms: conditions — Agnosia | interventions — Lidocaine; Magnesium Sulfate; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (L) (Active Comparator): Patients will receive lidocaine 3 mg/kg total of 40 ml (control group)
  Interventions: Drug: Lidocaine
- Group M (Active Comparator): Patients will receive lidocaine 3 mg/kg total of 40 ml plus Magnesium sulphate 30 mg/kg maximum 1.5 gm, mixed with the second 20 ml of block solution.
  Interventions: Drug: Magnesium Sulphate
- Group F (Active Comparator): Patients will receive lidocaine 3 mg/kg total of 40 ml plus fentanyl 1 mcg/kg, mixed with lidocaine given after the first 20 ml of block solution.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Lidocaine — Patients will receive lidocaine 3 mg/kg total of 40 ml (control group).
  Arms: Group (L)
Drug: Magnesium Sulphate — Patients will receive lidocaine 3 mg/kg total of 40 ml plus Magnesium sulphate 30 mg/kg maximum 1.5 gm, mixed with the second 20 ml of block solution.
  Arms: Group M
Drug: Fentanyl — Patients will receive lidocaine 3 mg/kg total of 40 ml plus fentanyl 1 mcg/kg, mixed with lidocaine given after the first 20 ml of block solution.
  Arms: Group F

SUMMARY:
Intravenous regional anesthesia is one of the well-known techniques of regional anesthesia for short surgical operations on the upper and lower limbs. It was first introduced back in 1908. Later on it was popularized even more for the same purpose by using two tourniquets to isolate an exsanguinated extremity then injection of local anesthesia. It was proved over time to be safe and effective with minimal side effects and complications.

Magnesium sulfate (MgSO4) has been used over the 20th century for prevention and treatment of pre-eclamptic and eclampsia seizures during pregnancy because of its superior safety profile over other drugs used for the same purpose. The specific mechanisms of action of magnesium sulfate still unclear but are probably multi-factorial. It may act as a vasodilator on peripheral as well as cerebral vasculature, to decrease peripheral vascular resistance and/or relieve vasoconstriction. Additionally, it may also protect the blood-brain barrier and limit cerebral edema formation, or it may also act as a central anticonvulsant.

Fentanyl; was first introduced back in 1990 for palliative use as fentanyl patch. Few years later, it became available in different forms of administration being highly lipophilic. Few years later it became the most widely used synthetic opioid in medicine. It is an opioid analgesic with a rapid onset and short duration of action. It is a potent μ-opioid receptor pure agonist. Fentanyl is 50 to 100 times more potent than morphine. Fentanyl has a relatively wide therapeutic index, which makes it a very safe surgical anesthetic drug when monitored carefully.

DETAILED DESCRIPTION:
Two Intravenous lines will be inserted one at a distal point on the arm to be blocked and other one in the other arm for fluids infusion. The block will be executed by injecting the target medicine in 10 ml increments in a blinded manner of total of 40 ml (study drugs diluted in normal saline 0.9% solution.

1. Group (L): will receive lidocaine 3 mg/kg total of 40 ml (control group)
2. Group (M): will receive lidocaine 3 mg/kg total of 40 ml plus Magnesium sulphate 30 mg/kg maximum 1.5 gm, mixed with the second 20 ml of block solution.
3. Group (F): will receive lidocaine 3 mg/kg total of 40 ml plus fentanyl 1 mcg/kg, mixed with lidocaine given after the first 20 ml of block solution.

Equipment: Local anesthetic agent: lidocaine HCl (2%), Rubber tourniquet, IV catheters (20- or 24-gauge), 500-mL or 1-L bag of IV solution (crystalloid), Infusion set, Pneumatic tourniquet, ideally with a double cuff, One Esmarch bandage (about 150 cm in length, 10 cm in width), Syringes.

Preparation: The patient lies in the supine position with the vein selected for block placement is readily accessible. Baseline vital signs are assessed; blood pressure, oxygen saturation, and ECG monitoring. Intravenous access in the non-operated extremity is obtained. Small doses of benzodiazepine for anxiolysis or small aliquots of opioids in case of discomfort will be available if needed. For safety and securing success, pneumatic cuffs will always be checked for air leaks prior to each IVRA procedure. Clinical staff performing the technique should have ready access to intra-lipid in case it is needed.

Technique:

1. Secure IV cannula in the extremity opposite to the block side.
2. A double pneumatic tourniquet is fixed on a padding layer of soft cloth or cotton with the proximal cuff high on the upper arm.
3. An IV cannula is inserted and secured into a peripheral vein of the operative limb, as far distally as possible.
4. The entire limb is elevated for 1 to 2 minutes to allow for passive exsanguination. Afterwards, while still keeping the limb high, a rubber (Esmarch) bandage is wrapped around it spirally from distal end proximally till the distal cuff of the double tourniquet.
5. The artery is digitally occluded by inflating the proximal cuff 100 mm Hg above systolic arterial blood pressure.
6. After reaching the correct pressure, the Esmarch bandage is removed.
7. A total of 40 mL of the study medicine according to the protocol is injected slowly in 10 ml increments via the IV catheter.
8. After the injection, the arm is lowered to the level of the table. The used IV cannula is removed, and in a sterile manner, pressure is quickly applied over the puncture site.

The onset of anesthesia is + 5 minutes after injection. When the patient reports the tourniquet pain, the distal cuff should be inflated and the proximal cuff is deflated about 20 to 30 minutes after the beginning of anesthesia

ELIGIBILITY:
Inclusion Criteria:

* scheduled for short surgical procedures (30 - 60 minutes) distal to elbow
* age 18-55 years old
* ASA I - II
* both genders
* average weight BMI (25 - 35).

Exclusion Criteria:

* seizure diseases
* allergy to the used medicine
* local infection
* patients with sickle cell anemia, Raynaud's disease, scleroderma, myasthenia gravis, significant cardiac or hepatic diseases.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
VAS score | 2 hours
  Onset of tourniquet pain after deflating proximal tourniquet. VAS consists of a straight line with the endpoints defining extreme limits WHERE 0='no pain AND 10= severe pain.

SECONDARY OUTCOMES:
3-point scale for motor function | 6 hours
  0: normal motor function, 1: reduced motor strength but able to move fingers, 2: complete motor block
3-point scale for sensory function | 6 hours
  0: normal sensation, 1: loss of sensation of cold (analgesia), 2: loss of sensation of touch (anesthesia).
Total Supplement Analgesia | 24 hours
  Total dose of pethidine 10 mg increments that will be used when the patients experience tourniquet pain >3 VAS.
Complications | 24 hours
  Number of patients with any intraoperative or postoperative complications will be recorded and treated.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No